CLINICAL TRIAL: NCT00883740
Title: Effects Of Pregabalin On Sleep Maintenance In Subjects With Fibromyalgia Syndrome And Sleep Maintenance Disturbance: A Randomized Placebo-Controlled 2-Way Crossover Polysomnography Study
Brief Title: Effects Of Pregabalin (Lyrica) On Sleep Maintenance In Subjects With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: A0081165
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2021-01-25 (Actual); Status verified 2011-07

CONDITIONS: Fibromyalgia; Sleep Disorders
Keywords: Fibromyalgia sleep maintenance disturbance pregabalin
MeSH Terms: conditions — Fibromyalgia; Sleep Wake Disorders | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Lyrica (Experimental): flexible dosing Lyrica 300-450mg/day
  Interventions: Drug: Pregabalin
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Pregabalin — Capsule, flexible dosing double-blind. Treatment duration is approximately 4 weeks titrated to 300-450 mg/day
  Arms: Lyrica
Drug: Placebo — Capsule, flexible dosing double-blind. Treatment duration is approximately 4 weeks
  Arms: Placebo

SUMMARY:
The purpose of the study is to demonstrate the effect of Lyrica on Wake after sleep onset in subjects with fibromyalgia with sleep maintenance disturbance (on polysomnogram)

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet diagnostic criteria for fibromyalgia;
* Subjects must report difficulty in maintaining sleep at least 3 times per week and meet Research Diagnostic Criteria (RDC) for insomnia disorder, corroborated by subject diary, and meet PSG inclusion criteria at visit 3.

Exclusion Criteria:

* History of active sleep disorder other than Research Diagnostic Criteria(RDC) insomnia criteria or any sleep or circadian rhythm disturbance;
* Use of medications known to affect sleep wake function by Visit 2;
* Involved in night or rotating shift work, or travel across >4 time zones 14 days prior to screening and during study; regular daytime napping
* PSG finding of apnea/hypopnea or periodic limb movement with arousal index >10/hr on either night of PSG.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 119 (Actual)
Dates: Start 2009-06; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (37):
- United States (25):
  - Pfizer Investigational Site, Phoenix, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Colorado Springs, Colorado
  - Pfizer Investigational Site, DeLand, Florida
  - Pfizer Investigational Site, Hallandale, Florida
  - Pfizer Investigational Site, Orange City, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, South Miami, Florida
  - Pfizer Investigational Site, Atlanta, Georgia
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Crestview Hills, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Baton Rouge, Louisiana
  - Pfizer Investigational Site, Hattiesburg, Mississippi
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Beachwood, Ohio
  - Pfizer Investigational Site, Cleveland, Ohio
  - Pfizer Investigational Site, Oklahoma City, Oklahoma
  - Pfizer Investigational Site, Duncansville, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Columbia, South Carolina
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
- Canada (7):
  - Pfizer Investigational Site, Calgary, Alberta
  - Pfizer Investigational Site, Edmonton, Alberta
  - Pfizer Investigational Site, Kelowna, British Columbia
  - Pfizer Investigational Site, Mississauga, Ontario
  - Pfizer Investigational Site, Point Edward, Ontario
  - Pfizer Investigational Site, Thornhill, Ontario
  - Pfizer Investigational Site, Toronto, Ontario
- Germany (5):
  - Pfizer Investigational Site, Berlin
  - Pfizer Investigational Site, Chemnitz
  - Pfizer Investigational Site, Göppingen
  - Pfizer Investigational Site, München
  - Pfizer Investigational Site, Schwerin

REFERENCES:
- [Derived] Roth T, Lankford DA, Bhadra P, Whalen E, Resnick EM. Effect of pregabalin on sleep in patients with fibromyalgia and sleep maintenance disturbance: a randomized, placebo-controlled, 2-way crossover polysomnography study. Arthritis Care Res (Hoboken). 2012 Apr;64(4):597-606. doi: 10.1002/acr.21595. PMID 22232085

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo, Then Pregabalin: Matching placebo twice daily in first intervention (treatment period 1, weeks 1-4) and pregabalin 75 milligrams (mg) up to 225 mg twice per day in second intervention (treatment period 2, weeks 7-10) after taper and washout period (weeks 5-6).
- Pregabalin, Then Placebo: Pregabalin 75 mg up to 225 mg twice per day in intervention (treatment period 1, weeks 1-4) and matching placebo twice daily in second intervention (treatment period 2, weeks 7-10) after taper and washout period (weeks 5-6).
Period: First Intervention
Arm/Group | Placebo, Then Pregabalin | Pregabalin, Then Placebo
Started | 60 | 59
Completed | 53 (1 participant not crossed to period 2 but continued on period 1, sponsor terminated as noncompliance) | 51
Not Completed | 7 | 8
Not completed — Lost to Follow-up | 1 | 0
Not completed — No longer willing to participate | 2 | 0
Not completed — Protocol Violation | 3 | 6
Not completed — Adverse Event | 1 | 2
Period: Taper and Washout Period (2 Weeks)
Arm/Group | Placebo, Then Pregabalin | Pregabalin, Then Placebo
Started | 54 (1 participant not crossed to period 2 but continued on period 1, sponsor terminated as noncompliance) | 51
Completed | 54 | 51
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Placebo, Then Pregabalin | Pregabalin, Then Placebo
Started | 53 (1 participant not crossed to period 2 but continued on period 1, sponsor terminated as noncompliance) | 51
Completed | 52 | 50
Not Completed | 1 | 1
Not completed — Protocol Violation | 1 | 0
Not completed — No longer willing to participate | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive matching placebo and Pregabalin, 75 up to 225 mg, twice per day in the first intervention and Pregabalin, 75 up to 225 mg, and matching placebo twice per day in the second intervention
Arm/Group | Entire Study Population
Number analyzed (Participants) | 119
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.4 (9.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103
  Male | 16
Medical Outcome Study Sleep Scale (MOS-SS) Sleep Disturbance Baseline Measure (Weeks 1 and 7) [Mean (Standard Deviation); unit: Scores on a Scale] — Sleep Disturbance subscale as measured by MOS-SS, a participant rated 12 item instrument. Baseline intervention period 1 collected at week 1 and baseline intervention period 2 collected at week 7. Scores were transformed and ranged from 0 to 100, higher scores indicated greater disturbance, negative changes indicated improvement.
  Scores on a Scale
    Week 1 Sleep Disturbance Placebo | 69.32 (17.48)
    Week 1 Sleep Disturbance Pregabalin | 69.29 (20.44)
    Week 7 Sleep Disturbance Placebo | 52.75 (24.77)
    Week 7 Sleep Disturbance Pregabalin | 51.51 (26.48)
MOS-SS Overall Sleep Index II Baseline Measure (Weeks 1 and 7) [Mean (Standard Deviation); unit: Scores on a Scale] — Overall Sleep Problem Index II determined by a 9 item index that provided a composite measure of overall sleep. Baseline intervention period 1 collected at week 1 and baseline intervention period 2 collected at week 7. Score ranged from 0 to 100, higher scores indicated greater sleep problems, negative changes indicated improvement.
  Scores on a Scale
    Week 1 Sleep Problems Index II Placebo | 62.82 (12.96)
    Week 1 Sleep Problems Index II Pregabalin | 63.21 (14.27)
    Week 7 Sleep Problems Index II Placebo | 47.22 (18.38)
    Week 7 Sleep Problems Index II Pregablin | 48.79 (19.89)

OUTCOME MEASURES:

1. Primary Outcome: Wake After Sleep Onset (WASO) at Weeks 5 and 11
Description: WASO was the sum of wake time during sleep measured in epochs (30 seconds of polysomnography [PSG]) recording) after the onset of persistent sleep and prior to final awakening and wake time after sleep (the number of epochs after the final awakening until the end of PSG recording [i.e. awake epoch immediately prior to the end of the recording]) on 2 consecutive nights divided by 2 at the end of each intervention period.
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or Early Termination (ET)
Population: Per Protocol Population (PP) = all randomized participants who received study medication at a dose of 300 or 450 mg/day and completed the study without any major protocol violations;
Measure: Least Squares Mean (Standard Error); unit: Minutes
Groups:
- Placebo: Matching Placebo administered twice daily in either first intervention treatment period 1, weeks 1-4 or second intervention treatment period 2, weeks 7-10.
- Pregabalin: Pregabalin administered twice daily in either first intervention treatment period 1, weeks 1-4 or second intervention treatment period 2, weeks 7-10.
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 83 | 83
Minutes | 70.69 (3.78) | 51.54 (3.78)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — P-value is based on a linear mixed effects model including sequence, period, and treatment as fixed factors and participant within sequence and within participant error as random factors; Mean Difference (Final Values) = -19.15, 95% CI 2-sided [-26.69 to -11.61]

2. Secondary Outcome: Wake Time During Sleep (WTDS)
Description: WTDS, as determined by PSG, was the total amount of time awake the participant experienced after the onset of persistent sleep and prior to the final awakening, or at the end of 8 hours of recording. WTDS was the sum of 2 consecutive nights of recordings divided by 2 at the end of each intervention period.
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or ET
Population: Intent to treat (ITT) population: randomized participants who received at least one dose of medication and had at least one efficacy evaluation
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Minutes | 63.38 (2.90) | 45.83 (2.93)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -17.54, 95% CI 2-sided [-23.29 to -11.80]

3. Secondary Outcome: Wake Time After Sleep (WTAS)
Description: WTAS, as determined by PSG, was the total amount of time awake after the final awakening until the end of the 8 hours. WTAS was the sum of 2 consecutive nights of recordings divided by 2 at the end of each intervention period.
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or ET
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Minutes | 9.19 (1.55) | 7.38 (1.57)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p = 0.3841, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.81, 95% CI 2-sided [-5.92 to 2.30]

4. Secondary Outcome: Total Sleep Time (TST)
Description: TST, as determined by PSG, was the number of non-wake epochs from the beginning of recording to the end of the recording. TST was the sum of 2 consecutive nights of recording divided by 2 at the end of each intervention period.
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or ET
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Minutes | 370.6 (4.65) | 396.2 (4.69)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 25.54, 95% CI 2-sided [17.48 to 33.61]

5. Secondary Outcome: Sleep Efficiency (SE)
Description: SE, as determined by PSG, was the TST divided by the time in bed, multiplied by 100. The sum of 2 consecutive nights of recording divided by 2 at the end of each intervention period.
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or ET
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Percentage of time asleep
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Percentage of time asleep | 77.21 (0.97) | 82.64 (0.98)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 5.42, 95% CI 2-sided [3.74 to 7.11]

6. Secondary Outcome: Number of Awakenings After Sleep Onset (NAASO 1)
Description: NAASO 1, as determined by PSG, was the number of times there was a wake period of at least one epoch in duration. Each entry counted was separated by a Stage 2 epoch, Stage 3 and 4 epoch, or Stage rapid eye movement (REM) epoch. The sum of 2 consecutive nights of recording was divided by 2 at the end of each intervention period.
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or ET
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Awakenings
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Awakenings | 26.92 (1.00) | 24.51 (1.00)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p = 0.0135, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.41, 95% CI 2-sided [-4.31 to -0.51]

7. Secondary Outcome: Number of Awakenings After Sleep Onset (NAASO 2)
Description: NAASO 2, as determined by PSG, was the number of times that there was a wake period of at least two epochs in duration. Each entry counted was separated by a Stage 2 epoch, Stage 3 and 4 epoch, or Stage REM epoch. The sum of 2 consecutive nights of recording divided by 2 at the end of each intervention period.
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or ET
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Awakenings
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Awakenings | 10.16 (0.44) | 8.63 (0.45)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p = 0.0008, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.53, 95% CI 2-sided [-2.41 to -0.66]

8. Secondary Outcome: Latency to Persistent Sleep (LPS)
Description: LPS, as determined by PSG, was the total number of epochs recorded on 2 consecutive nights divided by 2 at the end of each intervention period, from the beginning of the recording to the start of the first 20 consecutive non-wake epochs.
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or ET
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Minutes | 41.63 (3.70) | 34.45 (3.74)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p = 0.0447, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.18, 95% CI 2-sided [-14.18 to -0.17]

9. Secondary Outcome: WASO by Hour of the Night
Description: WASO, as determined by PSG, was the wake time during sleep (number of wake epochs after the onset of persistent sleep and prior to final awakening) and wake time after sleep (the number of epochs after the final awakening until the end of PSG recording) on 2 consecutive nights divided by 2 at the end of each intervention period by each individual hour (8 hours total).
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or ET
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Minutes
  Hour 1 | 1.96 (0.27) | 1.62 (0.28)
  Hour 2 | 5.66 (0.52) | 4.56 (0.53)
  Hour 3 | 7.09 (0.54) | 4.65 (0.55)
  Hour 4 | 8.95 (0.75) | 5.43 (0.75)
  Hour 5 | 10.55 (0.90) | 7.54 (0.90)
  Hour 6 | 11.26 (0.94) | 7.38 (0.95)
  Hour 7 | 10.96 (0.91) | 8.38 (0.92)
  Hour 8 | 17.08 (1.34) | 14.23 (1.35)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Hour 1; Test type: Superiority or Other; p = 0.3613, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.34, 95% CI 2-sided [-1.07 to 0.39]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Hour 2; Test type: Superiority or Other; p = 0.0686, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.10, 95% CI 2-sided [-2.29 to 0.09]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin; Hour 3; Test type: Superiority or Other; p = 0.0009, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.44, 95% CI 2-sided [-3.85 to -1.03]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin; Hour 4; Test type: Superiority or Other; p = 0.0002, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.52, 95% CI 2-sided [-5.33 to -1.71]
Statistical Analysis 5: Comparison: Placebo vs Pregabalin; Hour 5; Test type: Superiority or Other; p = 0.0065, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.01, 95% CI 2-sided [-5.16 to -0.86]
Statistical Analysis 6: Comparison: Placebo vs Pregabalin; Hour 6; Test type: Superiority or Other; p = 0.0024, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -3.89, 95% CI 2-sided [-6.36 to -1.41]
Statistical Analysis 7: Comparison: Placebo vs Pregabalin; Hour 7; Test type: Superiority or Other; p = 0.0366, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.59, 95% CI 2-sided [-5.01 to -0.16]
Statistical Analysis 8: Comparison: Placebo vs Pregabalin; Hour 8; Test type: Superiority or Other; p = 0.0593, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -2.85, 95% CI 2-sided [-5.82 to 0.11]

10. Secondary Outcome: WASO by Each Quarter of the Night
Description: WASO, as determined by PSG, was the sum of wake time during sleep (number of wake epochs after the onset of persistent sleep and prior to final awakening) and wake time after sleep (the number of epochs after the final awakening until the end of PSG recording) on 2 consecutive nights divided by 2 at the end of each intervention period by each individual quarter of the night (eight hours in 2 hour increments).
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or ET
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Minutes
  Quarter 1 | 7.23 (0.63) | 5.98 (0.64)
  Quarter 2 | 16.04 (1.05) | 10.04 (1.06)
  Quarter 3 | 21.73 (1.58) | 14.90 (1.60)
  Quarter 4 | 28.04 (1.98) | 22.60 (2.00)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Quarter 1; Test type: Superiority or Other; p = 0.1106, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -1.25, 95% CI 2-sided [-2.79 to 0.29]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Quarter 2; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.00, 95% CI 2-sided [-8.49 to -3.51]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin; Quarter 3; Test type: Superiority or Other; p = 0.0004, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.83, 95% CI 2-sided [-10.53 to -3.13]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin; Quarter 4; Test type: Superiority or Other; p = 0.0199, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.44, 95% CI 2-sided [-10.00 to -0.88]

11. Secondary Outcome: Slow Wave Sleep (SWS)
Description: SWS, as determined by PSG, Stage 3 plus 4 sleep divided by TST times 100 was the percentage of TST. The sum of 2 consecutive nights of recording divided by 2 at the end of each intervention period.
Time Frame: Week 5 (End of Intervention Period 1) and Week 11 (End of Intervention Period 2) or ET
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Percentage of total sleep time
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Percentage of total sleep time | 15.04 (1.01) | 17.18 (1.01)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Test type: Superiority or Other; p = 0.0024, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 2.14, 95% CI 2-sided [0.78 to 3.50]

12. Secondary Outcome: Change From Baseline in MOS-SS Sleep Disturbance at Weeks 5 and 11
Description: MOS-SS, a participant rated instrument used to assess sleep quantity and quality over the previous week, was comprised of 12 items yielding 7 subscale scores and 2 index composite index scores. Sleep Disturbance subscale score (4 items): individual scores were transformed (actual raw score minus lowest possible score divided by possible raw score range times 100) and ranged from 0 to 100; higher score indicated greater disturbance. Total score ranged=0 to 100; higher score indicates greater intensity of attribute. Change was score at week x minus score at baseline.
Time Frame: Week 1 (Baseline Intervention Period 1), Week 5 (End of Intervention Period 1), Week 7 (Baseline Intervention Period 2) and Week 11 (End of Intervention Period 2) or ET
Population: ITT; n: number of participants at specific time points
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Units on a scale
  Change Week 1 to Week 5 (n=59, 56) | -19.0 (2.98) | -27.1 (3.06)
  Change Week 7 to Week 11 (n=50, 52) | -2.23 (3.10) | -21.0 (3.04)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Week 5; Test type: Superiority or Other; p = 0.0591, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -8.13, 95% CI 2-sided [-16.59 to 0.32]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Week 11; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -18.81, 95% CI 2-sided [-27.43 to -10.20]

13. Secondary Outcome: Change From Baseline in MOS-SS Sleep Problems Index II Weeks 5 and 11
Description: MOS-SS, a participant rated instrument used to assess sleep quantity and quality over the previous week, was compromised of 12 items yielding 7 subscale scores and 2 index composite index scores. Composite index included Sleep Problems Index II (9 items), scores ranged from 0 to 100; higher scores indicated greater sleep problems. Change was score at week x minus score at baseline.
Time Frame: as for outcome 12
Population: ITT
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Units on a scale
  Change Week 1 to Week 5 (n=59, 56) | -16.4 (2.37) | -21.9 (2.43)
  Change Week 7 to Week 11 (50, 52) | -0.98 (2.51) | -14.4 (2.46)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Week 5; Test type: Superiority or Other; p = 0.1101, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.47, 95% CI 2-sided [-12.20 to 1.26]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Week 11; Test type: Superiority or Other; p = 0.0002, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.39, 95% CI 2-sided [-20.36 to -6.42]

14. Secondary Outcome: Sleep Quality
Description: Sleep Quality as meassured by numeric rating scale (NRS), a participant rated scale 0 to 10, (0 = very poor sleep, 10 = excellent sleep). Weekly values were calculated as the average of the participants daily diary scores.
Time Frame: Weeks 1, 2, 3 and 4 of Each Intervention Period or ET
Population: ITT; Last observation carried forward (LOCF)
Measure: Least Squares Mean (Standard Error); unit: Unit on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Unit on a scale
  Week 1 | 4.79 (0.16) | 5.70 (0.17)
  Week 2 | 4.95 (0.18) | 6.09 (0.18)
  Week 3 | 5.09 (0.17) | 5.96 (0.17)
  Week 4 | 5.17 (0.17) | 6.06 (0.17)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Week 1; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.91, 95% CI 2-sided [0.58 to 1.24]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Week 2; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 1.14, 95% CI 2-sided [0.76 to 1.53]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin; Week 3; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.87, 95% CI 2-sided [0.46 to 1.28]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin; Week 4; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.89, 95% CI 2-sided [0.51 to 1.26]

15. Secondary Outcome: Latency of Sleep Onset (LSO)
Description: LSO as reported on daily Subjective Sleep Questionnaire (SSQ), a participant reported subjective estimate of the amount of time to fall asleep after lights out. Weekly values were calculated as the average minutes reported on the participant's daily SSQ.
Time Frame: Weeks 1, 2, 3 and 4 of Each Intervention Period or ET
Population: ITT; LOCF
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Minutes
  Week 1 | 51.23 (2.61) | 43.56 (2.61)
  Week 2 | 49.94 (2.92) | 42.27 (2.92)
  Week 3 | 48.92 (4.01) | 43.24 (4.02)
  Week 4 | 46.70 (2.68) | 40.51 (2.68)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Week 1; Test type: Superiority or Other; p = 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.66, 95% CI 2-sided [-11.44 to -3.89]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Week 2; Test type: Superiority or Other; p = 0.0077, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -7.67, 95% CI 2-sided [-13.27 to -2.07]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin; Week 3; Test type: Superiority or Other; p = 0.2196, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -5.68, 95% CI 2-sided [-14.81 to 3.44]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin; Week 4; Test type: Superiority or Other; p = 0.0081, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -6.18, 95% CI 2-sided [-10.73 to -1.64]

16. Secondary Outcome: Daily Pain Score
Description: Pain intensity as measured by NRS; a participant rated scale 0 to 10 (0 = no pain to 10 = worst pain possible). Weekly values were calculated as the average of the participants daily pain scores.
Time Frame: Daily up to Day 73 or ET
Population: ITT; LOCF
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Units on a scale
  Week 1 | 6.12 (0.18) | 5.42 (0.18)
  Week 2 | 5.81 (0.18) | 5.10 (0.18)
  Week 3 | 5.73 (0.19) | 5.14 (0.19)
  Week 4 | 5.44 (0.20) | 4.92 (0.20)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Week 1; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.02 to -0.37]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Week 2; Test type: Superiority or Other; p = 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.06 to -0.36]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin; Week 3; Test type: Superiority or Other; p = 0.0014, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.59, 95% CI 2-sided [-0.95 to -0.24]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin; Week 4; Test type: Superiority or Other; p = 0.0084, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.90 to -0.14]

17. Secondary Outcome: Subjective Wake After Sleep Onset (sWASO)
Description: sWASO as reported on daily SSQ, a participant reported subjective estimate of the total amount of time the participant was awake after initial sleep onset until final awakening. Weekly values were calculated as the average of the participant's daily SSQ values.
Time Frame: Weeks 1, 2, 3 and 4 of Each Intervention Period or ET
Population: ITT; LOCF
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Minutes
  Week 1 | 80.86 (3.71) | 62.59 (3.73)
  Week 2 | 75.48 (3.91) | 59.43 (3.92)
  Week 3 | 74.97 (4.75) | 61.73 (4.76)
  Week 4 | 69.65 (4.20) | 59.40 (4.21)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Week 1; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -18.27, 95% CI 2-sided [-27.02 to -9.52]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Week 2; Test type: Superiority or Other; p = 0.0002, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -16.06, 95% CI 2-sided [-24.24 to -7.87]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin; Week 3; Test type: Superiority or Other; p = 0.0085, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -13.23, 95% CI 2-sided [-23.01 to -3.46]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin; Week 4; Test type: Superiority or Other; p = 0.0102, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -10.25, 95% CI 2-sided [-18.01 to -2.48]

18. Secondary Outcome: Subjective Total Sleep Time (sTST)
Description: sTST as reported on daily SSQ, a participant reported subjective estimate of the total amount of time the participant was asleep after lights out until final awakening. Weekly values were calculated as the average of the participants daily SSQ values.
Time Frame: Weeks 1, 2, 3 and 4 of Each Intervention Period or ET
Population: ITT; LOCF
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Placebo | Pregabalin
Number analyzed (Participants) | 109 | 108
Minutes
  Week 1 | 336.8 (5.40) | 361.7 (5.41)
  Week 2 | 341.9 (5.76) | 371.3 (5.77)
  Week 3 | 344.1 (5.73) | 370.9 (5.74)
  Week 4 | 352.5 (5.60) | 377.9 (5.61)
Statistical Analysis 1: Comparison: Placebo vs Pregabalin; Week 1; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 24.82, 95% CI 2-sided [13.25 to 36.40]
Statistical Analysis 2: Comparison: Placebo vs Pregabalin; Week 2; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 29.40, 95% CI 2-sided [18.59 to 40.21]
Statistical Analysis 3: Comparison: Placebo vs Pregabalin; Week 3; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 26.79, 95% CI 2-sided [15.37 to 38.21]
Statistical Analysis 4: Comparison: Placebo vs Pregabalin; Week 4; Test type: Superiority or Other; p < 0.0001, linear mixed effects model — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 25.44, 95% CI 2-sided [15.03 to 35.86]

ADVERSE EVENTS:
Description: The same event may appear as both an adverse events (AE) and a serious adverse events (SAE). However, what is presented are distinct events. An event may be categorized as serious in one participant and as nonserious in another participant, or one participant may have experienced both a serious and nonserious event during the study.
Arm/Group | Placebo | Pregabalin
Serious Adverse Events (participants affected / at risk) | 0/111 | 0/112
Other Adverse Events (participants affected / at risk) | 21/111 | 51/112
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=111) | Pregabalin (N=112)
nausea (Gastrointestinal disorders) | 3 | 8
dizziness (Nervous system disorders) | 11 | 34
headache (Nervous system disorders) | 9 | 10
somnolence (Nervous system disorders) | 5 | 23

LIMITATIONS AND CAVEATS:
The protocol specified analyses of secondary outcome measures (OMs) indicated OMs would use PP population; however all secondary OMs were analyzed using the ITT population in accordance with the statistical analysis plan.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.